CLINICAL TRIAL: NCT06498843
Title: Clinical Evaluation of the Effectiveness of Nasal Pump Spray Medical Devices DM004 and DM020 Based on Diluted Seawater in the Treatment of Colds, Rhinitis, Sinusitis, and Other Upper Respiratory Infections/Conditions
Brief Title: Efficacy of Two Nasal Products Based on Diluted Seawater in the Treatment of Upper Respiratory Infections/Conditions
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: YSLab (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUU524AA0972
Record Dates: First submitted 2024-06-27; First posted 2024-07-12 (Actual); Last update posted 2024-08-02 (Actual); Status verified 2024-07

CONDITIONS: Rhinitis; Sinusitis; Upper Respiratory Infections; Colds
MeSH Terms: conditions — Rhinitis; Sinusitis; Respiratory Tract Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- DM004-Isotonic nasal pump spray group (9g/L) (Experimental): Isotonic concentration. This solution has a concentration of mineral salts (concentration of halides expressed as NaCl: 9 g/L) similar to the human cells.
  Interventions: Other: administration of an isotonic seawater solution (9g/L) in the nose
- DM020-Hypertonic nasal pump spray group (21g/L) (Experimental): Hypertonic concentration. This solution has a concentration of mineral salts (concentration of halides expressed as NaCl: 21 g/L) higher than that of human cells.
  Interventions: Other: administration of a hypertonic seawater solution (21g/L) in the nose
- common practices (No Intervention): 1 control group with common practices people with an upper respiratory tract infection (cold, rhinitis, rhinopharyngitis...), not using nasal sprays nor nasal drops (in single-dose form, for example) but standard practices: hydration, rest, paracetamol if necessary

INTERVENTIONS:
Other: administration of an isotonic seawater solution (9g/L) in the nose — 1. pump spray group : people with an upper respiratory tract infection (cold, rhinitis, rhinopharyngitis, and other upper respiratory infections/conditions).
  2. sprays per nostril, at least 2 times a day up to 6 times a day. For 7 days
  Arms: DM004-Isotonic nasal pump spray group (9g/L)
Other: administration of a hypertonic seawater solution (21g/L) in the nose — 1. pump spray group : people with an upper respiratory tract infection (cold, rhinitis, rhinopharyngitis and other upper respiratory infections/conditions).
  2. sprays per nostril, at least 2 times a day up to 6 times a day. For 7 days
  Arms: DM020-Hypertonic nasal pump spray group (21g/L)

SUMMARY:
The goal of this interventional clinical trial is to test the safety and efficacy of two medical devices in subjects aged from 3 months old for the treatment of colds, rhinitis, sinusitis, and other upper respiratory infections/conditions for 7 days.

DETAILED DESCRIPTION:
The main endpoint is a symptom score evaluation. Severity is evaluated using the Jackson scale, which includes 8 symptoms (nasal discharge, nasal congestion, sneezing, sore throat, cough, headache, discomfort, chills) rated as absent, mild, moderate, or severe by the physician/investigator, on Day 0, immediately after the first use, on Day 3, and on Day 7.

The clinical evaluation is also conducted by the ENT specialist using the CGI (Clinical Global Impression - 7-point scale) on Day 0, immediately after the first use, on Day 3, and on Day 7, and by patients using the PGI (Patient Global Impression - 7-point scale) every day.

Concomitant treatments, number and timing of daily use, and tolerance (adverse effects) will also be studied.

ELIGIBILITY:
Inclusion Criteria:

* Autonomous adult, or minor with the consent of their legal representative
* Adults and children from 3 months old
* Ability of the patient (for adults) or their legal representative (for children) to follow the instructions for product use
* Having signed a free and informed consent to participate in the study expressed by the patient (for adults) or by their legal representative (for children) after being informed by the doctor.
* Person with an upper respiratory tract infection (cold, rhinitis, rhinopharyngitis…) with symptoms of nasal congestion and nasal discharge of moderate to severe intensity (Jackson derived score (nasal congestion + nasal discharge) ≥ 4 on Day 0).
* Persons with symptoms that started no more than 48 hours before the first visit

Exclusion Criteria:

* Person not showing cold symptoms, particularly no nasal congestion (chronic dry rhinitis, or Jackson derived score (nasal congestion + nasal discharge) < 4 on Day 0).
* Person undergoing treatment with a cortisone derivative, mucolytic, or medication containing pseudoephedrine or a similar product acting on nasal congestion or having used such a product within the 3 days preceding inclusion.
* Person having used a nasal wash product within the 3 days preceding inclusion.
* Person whose ability to use the product daily and complete the daily follow-up diary is in doubt.
* Person refusing to sign the informed consent form prior to the study.
* Person participating or having participated in any other clinical study within the 30 days preceding the study.
* Person participating in any other clinical study.

Min Age: 3 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 91 (Estimated)
Dates: Start 2025-01 (Estimated); Primary Completion 2025-03 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Measurement of the severity of Upper Respiratory Tract Symptoms (due to common cold, rhinitis, nasopharyngitis) using the Jackson scale. | on Day 0, immediately after the first use, Day 3, and Day 7.
  The severity of 8 symptoms (nasal discharge, nasal congestion, sneezing, sore throat, cough, headache, discomfort, chills) will be measured by an ENT specialist using the Jackson scale, which ranges from 0 to 3 (0 : none, 1 : mild, 2 : moderate, 3 : severe). The results will be reported as overall scores in comparison to Day 0 (baseline) and relative to the control group.
Clinical global impression using a scale | on Day 0, immediately after the first use, Day 3, and Day 7
  This measure involves the clinical evaluation of the patient's condition by an ENT specialist using the Clinical Global Impression (CGI) scale, which utilizes a 7-point scale ((1: greatly improved; 2: moderately improved; 3: slightly improved; 4: unchanged; 5: slightly worsened; 6: moderately worsened; 7: greatly worsened).
Patient global impression using a scale | on Day 0, immediately after the first use, Day 3, and Day 7
  This measure captures the patient's overall impression of their condition as perceived by the patient themselves. This subjective assessment will be recorded using a standardized 7-point scale ((1: greatly improved; 2: moderately improved; 3: slightly improved; 4: unchanged; 5: slightly worsened; 6: moderately worsened; 7: greatly worsened)), allowing comparison of their current state to the beginning of treatment. This provides insights into the patient's personal perception of their health status and treatment efficacy throughout the study period.
Questionnaire on subject's satisfaction and use of devices | Day 7
  This measure involves the subject's daily self-assessment using a questionnaire. The questionnaire is designed to capture the subject's perceptions and expériences during the study period. Moreover, this questionnaire will allow us to record the number and time of daily use of the devices under study.
Concomitant treatments using a questionnaire | Immediately after the first use, Day 3, and Day 7
  This measure involves documenting any additional treatments or medications that participants may be receiving alongside the study intervention. It includes recording the types of treatments, their frequencies, durations, and any changes during the study period.
Collection of Side Effects Using a Questionnaire | Immediately after the first use, Day 3, and Day 7
  This measure involves the daily recording of side effects experienced by participants. Side effects will be systematically documented each day, providing a comprehensive overview of the frequency and severity of adverse events throughout the study period. The number of patient with side effects will be notified

IPD SHARING:
Plan to Share IPD: No